CLINICAL TRIAL: NCT02516709
Title: CivaString Registry for Prostate Cancer
Brief Title: Linear Source Registry for Prostate Cancer
Acronym: CaRePC
Status: Completed | Type: Observational
Sponsor: CivaTech Oncology (Industry)
Responsible Party: Sponsor
Other Study IDs: CT003
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood, serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Linear LDR Source — The Linear LDR source is a permanent interstitial brachytherapy implant containing palladium-103 sources for the treatment of prostate cancer.

SUMMARY:
Ongoing follow up for subjects implanted with the Linear Source String for prostate cancer.

DETAILED DESCRIPTION:
This registry is being conducted to provide long term analysis on the use of the linear Civastring source for prostate cancer. Prospective data collection will record and demonstrate biochemical response rates. Long term side effects and adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Plans to remain in care of enrolling physician for 5 years
* > 5 years life expectancy
* Signed informed consent
* Enrolled within 6 weeks of implant or within 365 days of prior implant

Exclusion Criteria:

* Not willing or able to comply with protocol visit schedule

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently indicated for brachytherapy, implanted with the linear LDR source for prostate cancer with a life expectancy greater than 5 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Biochemical Response Rate (PSA) | Up to 5 years

SECONDARY OUTCOMES:
Side Effects (IPSS, IIEF, RFAS score) | Up to 5 years
Adverse Events | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristy Perez, PhD, Study Director — CivaTech Oncology
Locations (3):
- United States (3):
  - Chicago Prostate Cancer Center, Chicago, Illinois
  - Manhattan Medical Researcch, New York, New York
  - Bon Secours DePaul Medical Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No